CLINICAL TRIAL: NCT03150082
Title: An Open-label, Randomised, Single-dose, Two-period Cross-over Study to Evaluate Bioequivalence of GR37547 Ciprofloxacin 500 mg Tablet Versus Ciprofloxacin 500 mg Tablet Reference Product in Healthy Adult Participants Under Fasting Conditions
Brief Title: Bioequivalence Study Between GR37547 500 Milligrams (mg) Tablet Versus Ciprofloxacin 500 mg Tablet Reference Product in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 205730
Record Dates: First submitted 2017-05-10; First posted 2017-05-11 (Actual); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-06

CONDITIONS: Infections, Bacterial
Keywords: GR37547; Cross-over; Bioequivalence; Ciprofloxacin
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Crossover assignment: Subjects will receive treatment in one of the two sequences; Treatment A (GR37547 tablet) followed by Treatment B (ciprofloxacin reference tablet) or vice versa separated by a washout period of at least 7 days and not more than 14 days.
Masking Description: This will be an open-label study. Hence, masking will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence: A/B (Experimental): Eligible subjects will be randomized to receive a single dose of Treatment A (GR37547 500 mg tablet) followed by Treatment B (ciprofloxacin 500 mg reference tablet) administered orally on Day 1 in each treatment period. The washout period will be of at least 7 days and not more than 14 days.
  Interventions: Drug: GR37547 tablet; Drug: Ciprofloxacin reference tablet
- Treatment sequence: B/A (Experimental): Eligible subjects will be randomized to receive a single dose of Treatment B (ciprofloxacin 500 mg reference tablet) followed by Treatment A (GR37547 500 mg tablet) administered orally. The washout period will be of at least 7 days and not more than 14 days.
  Interventions: Drug: GR37547 tablet; Drug: Ciprofloxacin reference tablet

INTERVENTIONS:
Drug: GR37547 tablet — A single tablet of GR37547 should be taken orally with 240 mL of water. GR37547 500 mg tablet will be a white to off white capsule shape with break line on upper side and embossed "GSK500"on lower side.
Drug: Ciprofloxacin reference tablet — A single tablet of ciprofloxacin reference should be taken orally with 240 mL of water. Ciprofloxacin 500 mg reference will be nearly white to slightly yellowish film coated oblong tablets with break line and ''CIP 500" marked on upper side and "BAYER" on lower side.

SUMMARY:
This two-period cross-over study will evaluate bioequivalence of GR37547 (ciprofloxacin 500 mg) tablet versus ciprofloxacin 500 mg reference tablet in healthy adult subjects under fasting conditions. Subjects will receive Treatment A (GR37547 tablet) and Treatment B (ciprofloxacin reference tablet) in crossover manner, separated by a washout period of at least 7 days and not more than 14 days. The total duration of study for each subject will be approximately 5-7 weeks. This study will enroll approximately 26 healthy adult subjects at a single center.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* Healthy, non-smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required,agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19-30 kg per meter square (kg/m^2) (inclusive).
* Healthy Male or female subjects: Male subjects: A male subject must agree to use contraception during the treatment period and for at least 5 days, after the last dose of study treatment and refrain from donating sperm during this period; Female subjects: A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study treatment.
* The investigator is responsible for ensuring that male and female study subjects understand how to correctly use the methods of contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neuromuscular, psychiatric, auto-immune or neurological disorders.
* History of convulsions.
* Any other condition that is capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* History of any malignancies or chemotherapy/radiation within the past 5 years excluding treated squamous carcinoma of the skin and adequately excised basal cell carcinoma.
* History of kidney, heart or lung transplants.
* History or presence of rheumatoid arthritis.
* Presence of hypocalcaemia where the serum potassium is < lower limit of normal (LLN).
* Presence of hypomagnesaemia where the serum magnesium is < LLN.
* Fasting blood glucose >=7 millimoles (mmol)/liter (L).
* Serum glucose-6-phosphate dehydrogenase < LLN.
* Abnormal renal function, as determined by creatinine clearance and considered as clinically significant by the investigator will be excluded.
* Alanine transaminase (ALT) >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Excessive alkalinity of the urine (potential of hydrogen [pH] >=9), as determined on Day -1.
* Abnormal BP as determined by the investigator.
* QT interval corrected for heart rate according to Bazett's formula (QTcB) >450 milliseconds (msec). Subjects with a known risk of QT prolongation will be excluded. For purposes of data analysis, only QTcB, will be used
* Past or intended use of over-the-counter or prescription medication including herbal medications, within 14 days prior to dosing unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.
* Where participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 90 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation within the last 90 days before signing of consent in this or any other clinical study involving an investigational study treatment.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or a Positive Hepatitis C antibody test result at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy including allergy to quinolones that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 6 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, randomized, single-dose, two-period cross-over study to evaluate bioequivalence of GR37547 ciprofloxacin 500 milligrams (mg) test product versus ciprofloxacin 500 mg reference product in healthy adult participants under fasting conditions. Participants were enrolled at a single center in South Africa.
Pre-assignment Details: Participants received treatment in one of the two sequences; Treatment A (GR37547) followed by Treatment B (ciprofloxacin reference) or vice versa in each of the treatment period 1 and 2. A total number of 26 participants were randomized.
Groups:
- GR37547 Followed by Ciprofloxacin Reference Product: Eligible participants received a single dose of Treatment A (GR37547 500 mg tablet), administered orally on Day 1 in treatment period 1. It was followed by a washout period of at least 7 days and not more than 14 days. Participants received Treatment B (ciprofloxacin 500 mg reference tablet), administered orally on Day 1 in treatment period 2.
- Ciprofloxacin Reference Product Followed by GR37547: Eligible participants received Treatment B (ciprofloxacin 500 mg reference tablet), administered orally on Day 1 in treatment period 1. It was followed by a washout period of at least 7 days and not more than 14 days. Participants received a single dose of Treatment A (GR37547 500 mg tablet), administered orally on Day 1 in treatment period 2.
Period: Treatment Period 1 (Up to 4 Weeks)
Arm/Group | GR37547 Followed by Ciprofloxacin Reference Product | Ciprofloxacin Reference Product Followed by GR37547
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout Period (Up to 4 Weeks)
Arm/Group | GR37547 Followed by Ciprofloxacin Reference Product | Ciprofloxacin Reference Product Followed by GR37547
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Treatment Period 2 (Up to 4 Weeks)
Arm/Group | GR37547 Followed by Ciprofloxacin Reference Product | Ciprofloxacin Reference Product Followed by GR37547
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Eligible participants received a single dose of Treatment A (GR37547 500 mg tablet) followed by Treatment B (ciprofloxacin 500 mg reference tablet) or vice versa, administered orally on Day 1 in each treatment period 1 and 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.5 (5.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 18
  White -White/Caucasian/European Heritage | 6
  Other-Mixed Race | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration Within a Participant Across All Treatments (AUC[0-t]) for Ciprofloxacin
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of ciprofloxacin under fasted state. Pharmacokinetic analysis of ciprofloxacin was conducted using non-compartmental methods. Pharmacokinetic Population comprised of participants who completed the study and for whom primary pharmacokinetic parameters could be calculated for all treatment periods were included in the statistical pharmacokinetic analysis of the study.
Time Frame: Pre-dose and 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 3.50, 4.50, 6.00, 8.00, 12.00, 18.00 hours post-dose on Day 1; 24.00 hours post-dose on Day 2 in each treatment period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Groups:
- Ciprofloxacin 500 mg Reference: Eligible participants received ciprofloxacin 500 mg tablet reference product (Treatment B) , administered orally on Day 1 in each treatment period 1 and 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
- GR37547 500 mg: Eligible participants received GR37547 ciprofloxacin 500 mg tablet test product (Treatment A), administered orally on Day 1 in each treatment period 1 and 2. The washout period was of at least 7 days and not more than 14 days between the treatment periods.
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Hour*nanogram per milliliter | 11600 (22.5) | 11300 (27.7)
Statistical Analysis 1: Comparison: Ciprofloxacin 500 mg Reference vs GR37547 500 mg; Test type: Equivalence — Bio-equivalence analysis comparing ciprofloxacin test and reference product has been presented; Percent ratio = 96.88, 90% CI 2-sided [91.13 to 103.00] — Percent ratio (GR37547 500 mg/ciprofloxacin 500 mg reference) has been presented

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ciprofloxacin
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of ciprofloxacin under fasted state. Pharmacokinetic analysis of ciprofloxacin was conducted using non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Nanogram per milliliter | 3140 (21.6) | 2940 (29.6)
Statistical Analysis 1: Comparison: Ciprofloxacin 500 mg Reference vs GR37547 500 mg; Test type: Equivalence — Bio-equivalence analysis comparing ciprofloxacin test and reference product has been presented; Percent ratio = 93.16, 90% CI 2-sided [86.09 to 100.82] — Percent ratio (GR37547 500 mg/ciprofloxacin 500 mg reference) has been presented

3. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) for Ciprofloxacin
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Hour*nanogram per milliliter | 12000 (22.0) | 11600 (27.3)
Statistical Analysis 1: Comparison: Ciprofloxacin 500 mg Reference vs GR37547 500 mg; Test type: Equivalence — Bio-equivalence analysis comparing ciprofloxacin test and reference product has been presented; Percent ratio = 96.96, 90% CI 2-sided [91.17 to 103.11] — Percent ratio (GR37547 500 mg/ciprofloxacin 500 mg reference) has been presented

4. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for Ciprofloxacin
Description: Blood samples were collected from participants at indicated time points in each of the treatment period 1 and 2, after administration of study treatment to investigate the pharmacokinetics of ciprofloxacin under fasted state. Pharmacokinetic analysis of ciprofloxacin was conducted using non-compartmental methods. Tmax of ciprofloxacin was analyzed using a nonparametric test to compute point estimate of the median and full range.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Hours | 1.253 [0.50 to 2.00] | 1.009 [0.50 to 2.52]
Statistical Analysis 1: Comparison: Ciprofloxacin 500 mg Reference vs GR37547 500 mg; Test type: Equivalence — Bio-equivalence analysis comparing ciprofloxacin test and reference product has been presented; p = 0.3499, Wilcoxon signed-rank test — P value was analyzed using a nonparametric "Wilcoxon signed-rank test"

5. Secondary Outcome: Percentage of AUC (0-infinity) Obtained by Extrapolation (Percentage AUCex) for Ciprofloxacin
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUCex
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Percentage of AUCex | 2.83 (31.6) | 2.85 (36.9)

6. Secondary Outcome: Terminal Phase Half-life (t1/2) for Ciprofloxacin
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Ciprofloxacin 500 mg Reference | GR37547 500 mg
Number analyzed (Participants) | 25 | 25
Hours | 5.02 (13.5) | 4.82 (19.8)

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious AEs (Non-SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, is a congenital anomaly/ birth defect or other situations. The analysis was performed on Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment. Participants were analyzed according to the treatment they actually received.
Time Frame: Up to 4 weeks in each treatment period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Participants
  Any Non-SAE | 6 | 6
  Any SAE | 0 | 0

8. Secondary Outcome: Alanine Aminotransferase (ALT), Alkaline Phosphatase (Alk Phos), Aspartate Aminotransferase (AST) and Lactate Dehydrogenase (LD) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including ALT, Alk phos, AST and LD. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Units per liter
  ALT; Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  ALT; Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 17.3 (10.50) | 18.0 (10.85)
  ALT; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  ALT; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 15.3 (8.74) | 16.4 (12.71)
  ALT; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  ALT; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 21.2 (22.95) | 16.6 (10.75)
  ALT; Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  ALT; Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 20.8 (28.51) | 14.6 (9.41)
  Alk Phos;Period 1;Day -1,24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Alk Phos;Period 1;Day -1,24 Hours Pre-dose;n=13,13 | 72.7 (21.83) | 65.5 (15.69)
  Alk Phos;Period 1;Day 2,24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Alk Phos;Period 1;Day 2,24 Hours Post-dose;n=13,13 | 67.6 (22.88) | 61.0 (15.02)
  Alk Phos;Period 2;Day -1,24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Alk Phos;Period 2;Day -1,24 Hours Pre-dose;n=13,12 | 63.8 (15.66) | 74.9 (22.51)
  Alk Phos;Period 2;Day 2,24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Alk Phos;Period 2;Day 2,24 Hours Post-dose;n=13,12 | 59.4 (13.48) | 70.3 (23.59)
  AST; Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  AST; Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 21.3 (6.82) | 20.8 (3.39)
  AST; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  AST; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 18.2 (4.51) | 17.5 (3.67)
  AST; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  AST; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 22.6 (8.83) | 21.2 (8.79)
  AST; Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  AST; Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 19.4 (7.40) | 18.3 (5.73)
  LD; Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  LD; Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 324.9 (57.56) | 322.2 (56.71)
  LD; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  LD; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 280.6 (47.22) | 273.9 (46.00)
  LD; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  LD; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 331.4 (49.08) | 327.0 (54.87)
  LD; Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  LD; Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 287.2 (52.27) | 291.8 (43.00)

9. Secondary Outcome: Blood Urea Nitrogen (BUN) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of BUN. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Milligrams per deciliter
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 11.322 (3.810) | 10.392 (2.201)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 10.909 (2.611) | 10.073 (1.510)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 11.444 (3.133) | 11.682 (2.241)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 10.548 (1.674) | 11.583 (1.860)

10. Secondary Outcome: Calcium, Chloride, Glucose, Magnesium, Potassium and Sodium at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including calcium, chloride, glucose, magnesium, potassium and sodium. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Millimoles per liter
  Calcium;Period 1;Day -1,24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Calcium;Period 1;Day -1,24 Hours Pre-dose;n=13,13 | 2.354 (0.072) | 2.337 (0.088)
  Calcium;Period 1;Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Calcium;Period 1;Day 2, 24 Hours Post-dose;n=13,13 | 2.269 (0.082) | 2.250 (0.081)
  Calcium;Period 2;Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Calcium;Period 2;Day -1, 24 Hours Pre-dose;n=13,12 | 2.335 (0.103) | 2.348 (0.059)
  Calcium;Period 2;Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Calcium;Period 2;Day 2, 24 Hours Post-dose;n=13,12 | 2.265 (0.069) | 2.309 (0.076)
  Chloride;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Chloride;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 104.41 (2.077) | 104.38 (1.305)
  Chloride;Period 1;Day 2,24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Chloride;Period 1;Day 2,24 Hours Post-dose;n=13,13 | 106.29 (1.715) | 106.68 (1.392)
  Chloride;Period 2;Day -1,24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Chloride;Period 2;Day -1,24 Hours Pre-dose;n=13,12 | 103.65 (1.975) | 103.74 (1.641)
  Chloride;Period 2;Day 2,24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Chloride;Period 2;Day 2,24 Hours Post-dose;n=13,12 | 107.22 (1.213) | 106.68 (1.471)
  Glucose;Period 1; Day -1,24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Glucose;Period 1; Day -1,24 Hours Pre-dose;n=13,13 | 4.691 (0.260) | 4.666 (0.312)
  Glucose;Period 1; Day 2,24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Glucose;Period 1; Day 2,24 Hours Post-dose;n=13,13 | 4.738 (0.272) | 4.669 (0.191)
  Glucose;Period 2;Day -1,24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Glucose;Period 2;Day -1,24 Hours Pre-dose;n=13,12 | 4.377 (0.238) | 4.696 (0.381)
  Glucose;Period 2;Day 2,24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Glucose;Period 2;Day 2,24 Hours Post-dose;n=13,12 | 4.508 (0.235) | 4.608 (0.255)
  Magnesium;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Magnesium;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 0.830 (0.052) | 0.823 (0.043)
  Magnesium;Period 1;Day2, 24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Magnesium;Period 1;Day2, 24Hours Post-dose;n=13,13 | 0.813 (0.054) | 0.828 (0.039)
  Magnesium;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Magnesium;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 0.800 (0.055) | 0.809 (0.075)
  Magnesium;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Magnesium;Period 2;Day 2,24Hours Post-dose;n=13,12 | 0.836 (0.048) | 0.841 (0.048)
  Potassium;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Potassium;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 4.431 (0.335) | 4.450 (0.251)
  Potassium;Period 1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Potassium;Period 1;Day 2,24Hours Post-dose;n=13,13 | 4.511 (0.283) | 4.349 (0.248)
  Potassium;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Potassium;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 4.518 (0.339) | 4.581 (0.317)
  Potassium;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Potassium;Period 2;Day 2,24Hours Post-dose;n=13,12 | 4.341 (0.218) | 4.570 (0.338)
  Sodium;Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Sodium;Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 140.15 (2.304) | 139.85 (2.478)
  Sodium; Period 1;Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Sodium; Period 1;Day 2, 24 Hours Post-dose;n=13,13 | 141.46 (1.506) | 141.62 (1.502)
  Sodium;Period 2; Day -1,24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Sodium;Period 2; Day -1,24 Hours Pre-dose;n=13,12 | 138.54 (1.561) | 139.00 (1.809)
  Sodium; Period 2;Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Sodium; Period 2;Day 2, 24 Hours Post-dose;n=13,12 | 140.62 (1.325) | 140.92 (1.443)

11. Secondary Outcome: Total Bilirubin (Total Bil), Direct Bilirubin (Direct Bil) and Creatinine (Creat) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of clinical chemistry parameters including total bil, direct bil and creat. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Moles per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Moles per liter
  Total bil;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Total bil;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 9.39 (2.415) | 9.05 (5.429)
  Total bil;Period 1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Total bil;Period 1;Day 2,24Hours Post-dose;n=13,13 | 8.18 (3.176) | 7.88 (4.556)
  Total bil;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Total bil;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 9.29 (5.012) | 8.78 (4.888)
  Total bil;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Total bil;Period 2;Day 2,24Hours Post-dose;n=13,12 | 8.10 (4.383) | 6.90 (3.207)
  Direct bil;Period 1;Day-1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Direct bil;Period 1;Day-1,24Hours Pre-dose;n=13,13 | 3.89 (0.779) | 3.46 (1.693)
  Direct bil;Period 1;Day2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Direct bil;Period 1;Day2,24Hours Post-dose;n=13,13 | 3.14 (0.965) | 2.87 (1.297)
  Direct bil;Period2;Day-1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Direct bil;Period2;Day-1,24Hours Pre-dose;n=13,12 | 3.50 (1.477) | 3.40 (1.285)
  Direct bil;Period2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Direct bil;Period2;Day 2,24Hours Post-dose;n=13,12 | 3.12 (1.336) | 2.90 (0.932)
  Creat; Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Creat; Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 76.3 (11.24) | 72.2 (17.22)
  Creat; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Creat; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 79.2 (12.33) | 75.2 (18.15)
  Creat; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Creat; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 71.6 (15.61) | 74.8 (13.13)
  Creat Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Creat Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 73.4 (17.16) | 76.8 (12.62)

12. Secondary Outcome: Total Protein at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for the analysis of total Protein. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Grams per liter
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 75.45 (5.090) | 74.58 (3.093)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 70.32 (5.023) | 68.82 (4.013)
  Period 2; Day -1, 24 Hours Pre-dose ;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose ;n=13,12 | 73.31 (4.296) | 76.51 (4.268)
  Period 2; Day 2, 24 Hours Post-dose ;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose ;n=13,12 | 70.23 (2.985) | 72.06 (2.831)

13. Secondary Outcome: Platelets, Neutrophils, Monocytes, Lymphocytes, Leucocyte, Eosinophils and Basophils at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematology parameters including platelets, neutrophils, monocytes, lymphocytes, leucocyte, eosinophils and basophils. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
10^9 cells per liter
  Basophils;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Basophils;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 0.032 (0.020) | 0.022 (0.012)
  Basophils;Period1; Day2,24Hours Post-dose ;n=13,13: number analyzed (Participants) | 13 | 13
  Basophils;Period1; Day2,24Hours Post-dose ;n=13,13 | 0.031 (0.019) | 0.018 (0.011)
  Basophils;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Basophils;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 0.019 (0.012) | 0.033 (0.019)
  Basophils;Period 2;Day2, 24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Basophils;Period 2;Day2, 24Hours Post-dose;n=13,12 | 0.019 (0.010) | 0.031 (0.021)
  Eosinophils;Period1;Day-1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Eosinophils;Period1;Day-1,24Hours Pre-dose;n=13,13 | 0.237 (0.259) | 0.132 (0.071)
  Eosinophils;Period1;Day2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Eosinophils;Period1;Day2,24Hours Post-dose;n=13,13 | 0.209 (0.186) | 0.128 (0.060)
  Eosinophils;Period2;Day-1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Eosinophils;Period2;Day-1,24Hours Pre-dose;n=13,12 | 0.127 (0.068) | 0.286 (0.259)
  Eosinophils;Period2;Day2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Eosinophils;Period2;Day2,24Hours Post-dose;n=13,12 | 0.115 (0.073) | 0.286 (0.271)
  Leucocyte;Period 1;Day-1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Leucocyte;Period 1;Day-1,24Hours Pre-dose;n=13,13 | 5.247 (1.509) | 5.915 (1.473)
  Leucocyte;Period 1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Leucocyte;Period 1;Day 2,24Hours Post-dose;n=13,13 | 4.897 (1.232) | 5.269 (1.349)
  Leucocyte;Period 2;Day-1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Leucocyte;Period 2;Day-1,24Hours Pre-dose;n=13,12 | 6.373 (1.577) | 5.508 (1.246)
  Leucocyte;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Leucocyte;Period 2;Day 2,24Hours Post-dose;n=13,12 | 5.118 (1.159) | 4.973 (0.797)
  Lymphocytes;Period1;Day -1,24Hours Predose;n=13,13: number analyzed (Participants) | 13 | 13
  Lymphocytes;Period1;Day -1,24Hours Predose;n=13,13 | 1.885 (0.430) | 2.215 (0.596)
  Lymphocytes;Period1;Day2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Lymphocytes;Period1;Day2,24Hours Post-dose;n=13,13 | 1.781 (0.379) | 2.026 (0.555)
  Lymphocytes;Period2;Day -1,24Hours Predose;n=13,12: number analyzed (Participants) | 13 | 12
  Lymphocytes;Period2;Day -1,24Hours Predose;n=13,12 | 2.567 (0.641) | 2.201 (0.470)
  Lymphocytes;Period2;Day2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Lymphocytes;Period2;Day2,24Hours Post-dose;n=13,12 | 1.938 (0.451) | 1.883 (0.310)
  Monocytes;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Monocytes;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 0.471 (0.176) | 0.535 (0.124)
  Monocytes;Period 1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Monocytes;Period 1;Day 2,24Hours Post-dose;n=13,13 | 0.452 (0.157) | 0.495 (0.156)
  Monocytes;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Monocytes;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 0.560 (0.167) | 0.519 (0.166)
  Monocytes;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Monocytes;Period 2;Day 2,24Hours Post-dose;n=13,12 | 0.451 (0.134) | 0.443 (0.153)
  Neutrophil;Period1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Neutrophil;Period1;Day -1,24Hours Pre-dose;n=13,13 | 2.622 (1.130) | 3.012 (1.225)
  Neutrophil;Period1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Neutrophil;Period1;Day 2,24Hours Post-dose;n=13,13 | 2.424 (1.393) | 2.602 (1.226)
  Neutrophil;Period2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Neutrophil;Period2;Day -1,24Hours Pre-dose;n=13,12 | 3.100 (1.154) | 2.469 (0.774)
  Neutrophil;Period2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Neutrophil;Period2;Day 2,24Hours Post-dose;n=13,12 | 2.594 (0.802) | 2.330 (0.575)
  Platelets;Period 1;Day -1,24Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Platelets;Period 1;Day -1,24Hours Pre-dose;n=13,13 | 313.4 (62.52) | 292.5 (71.81)
  Platelets;Period 1;Day 2,24Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Platelets;Period 1;Day 2,24Hours Post-dose;n=13,13 | 295.1 (63.24) | 281.5 (62.29)
  Platelets;Period 2;Day -1,24Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Platelets;Period 2;Day -1,24Hours Pre-dose;n=13,12 | 307.6 (70.01) | 325.2 (77.79)
  Platelets;Period 2;Day 2,24Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Platelets;Period 2;Day 2,24Hours Post-dose;n=13,12 | 296.5 (72.54) | 299.9 (65.97)

14. Secondary Outcome: Mean Corpuscular Volume (MCV) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of MCV. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Femtoliter
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 82.95 (4.668) | 83.01 (4.613)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 82.88 (4.735) | 82.65 (4.406)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 83.42 (4.511) | 83.30 (4.657)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 83.21 (4.397) | 83.27 (4.660)

15. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of MCH. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Picogram
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 29.05 (2.172) | 28.86 (1.809)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 29.13 (2.240) | 29.02 (1.940)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 28.89 (1.870) | 28.88 (2.316)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 28.94 (1.829) | 29.00 (2.324)

16. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC) and Hemoglobin (Hb) at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematology parameters including MCHC and Hb. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per deciliter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Grams per deciliter
  MCHC;Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  MCHC;Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 35.00 (1.078) | 34.78 (0.829)
  MCHC;Period 1; Day 2, 24 Hours Post-dose; n=13,13: number analyzed (Participants) | 13 | 13
  MCHC;Period 1; Day 2, 24 Hours Post-dose; n=13,13 | 35.12 (1.083) | 35.09 (0.852)
  MCHC; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  MCHC; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 34.62 (0.873) | 34.58 (1.245)
  MCHC;Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  MCHC;Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 34.78 (0.755) | 34.78 (1.176)
  Hb; Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Hb; Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 14.48 (1.862) | 14.20 (1.469)
  Hb; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Hb; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 14.04 (1.782) | 13.74 (1.669)
  Hb; Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Hb; Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 13.88 (1.499) | 14.23 (2.119)
  Hb; Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Hb; Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 13.41 (1.574) | 13.82 (1.985)

17. Secondary Outcome: Percent Reticulocytes at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of percent reticulocytes. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Percentage of reticulocytes
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 2.277 (0.442) | 2.069 (0.250)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 2.085 (0.369) | 2.123 (0.280)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 2.362 (0.275) | 2.167 (0.347)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 0.931 (0.155) | 1.883 (0.513)

18. Secondary Outcome: Hematocrit at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of hematocrit. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Proportion of red blood cells in blood
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 0.413 (0.044) | 0.408 (0.036)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 0.399 (0.041) | 0.391 (0.041)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 0.400 (0.035) | 0.410 (0.051)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 0.385 (0.040) | 0.396 (0.047)

19. Secondary Outcome: Erythrocyte Count at Indicated Time-points
Description: Blood samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2 for evaluation of erythrocyte count. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
10^12 cells per liter
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day -1, 24 Hours Pre-dose;n=13,13 | 4.975 (0.415) | 4.922 (0.442)
  Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 4.812 (0.429) | 4.733 (0.466)
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day -1, 24 Hours Pre-dose;n=13,12 | 4.804 (0.403) | 4.918 (0.498)
  Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 4.630 (0.441) | 4.752 (0.454)

20. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for Urinalysis
Description: Urine samples were collected from participants on Day -1 and Day 2 of each treatment period 1 and 2. The number of participants with abnormal (clinically significant) findings for urinalysis have been presented.
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for Electrocardiogram (ECG) Parameters
Description: A single 12-lead ECGs was obtained on Day 1 and Day 2 of each treatment period 1 and 2 using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT corrected (QTc) intervals. The number of participants with abnormal (clinically significant) findings for ECG parameters have been presented.
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

22. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Indicated Time-points
Description: Blood pressure of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Millimeters of mercury
  SBP;Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  SBP;Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13 | 107.2 (9.81) | 109.8 (9.25)
  SBP;Period 1; Day 1, 2 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  SBP;Period 1; Day 1, 2 Hours Post-dose;n=13,13 | 108.4 (9.11) | 106.3 (9.68)
  SBP;Period 1; Day 1, 4 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  SBP;Period 1; Day 1, 4 Hours Post-dose;n=13,13 | 109.2 (10.49) | 108.8 (7.22)
  SBP;Period 1; Day 1, 6 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  SBP;Period 1; Day 1, 6 Hours Post-dose;n=13,13 | 106.3 (9.36) | 104.1 (7.76)
  SBP;Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  SBP;Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 104.6 (8.83) | 105.5 (6.29)
  SBP;Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  SBP;Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12 | 104.0 (5.83) | 105.8 (4.83)
  SBP;Period 2; Day 1, 2 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  SBP;Period 2; Day 1, 2 Hours Post-dose;n=13,12 | 106.9 (5.82) | 104.9 (9.67)
  SBP;Period 2; Day 1, 4 Hours Post-dose=13,12: number analyzed (Participants) | 13 | 12
  SBP;Period 2; Day 1, 4 Hours Post-dose=13,12 | 105.0 (7.60) | 108.9 (8.02)
  SBP;Period 2; Day 1, 6 Hours Post-dose=13,12: number analyzed (Participants) | 13 | 12
  SBP;Period 2; Day 1, 6 Hours Post-dose=13,12 | 103.6 (9.18) | 107.8 (7.56)
  SBP;Period 2; Day 2, 24 Hours Post-dose=13,12: number analyzed (Participants) | 13 | 12
  SBP;Period 2; Day 2, 24 Hours Post-dose=13,12 | 109.1 (5.91) | 107.5 (6.88)
  DBP;Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  DBP;Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13 | 60.5 (8.75) | 62.6 (7.46)
  DBP;Period 1; Day 1, 2 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  DBP;Period 1; Day 1, 2 Hours Post-dose;n=13,13 | 60.0 (5.76) | 61.2 (7.18)
  DBP; Period 1;Day 1, 4 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  DBP; Period 1;Day 1, 4 Hours Post-dose;n=13,13 | 60.2 (6.89) | 59.8 (5.64)
  DBP; Period 1;Day 1, 6 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  DBP; Period 1;Day 1, 6 Hours Post-dose;n=13,13 | 56.2 (6.38) | 56.5 (3.62)
  DBP; Period 1; Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  DBP; Period 1; Day 2, 24 Hours Post-dose;n=13,13 | 59.1 (4.92) | 60.5 (6.81)
  DBP;Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  DBP;Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12 | 60.7 (6.14) | 60.0 (4.00)
  DBP;Period 2; Day 1, 2 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  DBP;Period 2; Day 1, 2 Hours Post-dose;n=13,12 | 60.8 (3.87) | 59.7 (6.69)
  DBP; Period 2;Day 1, 4 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  DBP; Period 2;Day 1, 4 Hours Post-dose;n=13,12 | 57.7 (5.63) | 60.9 (4.96)
  DBP; Period 2;Day 1, 6 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  DBP; Period 2;Day 1, 6 Hours Post-dose;n=13,12 | 55.2 (3.39) | 56.5 (3.92)
  DBP; Period 2; Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  DBP; Period 2; Day 2, 24 Hours Post-dose;n=13,12 | 64.5 (5.98) | 60.8 (4.53)

23. Secondary Outcome: Respiratory Rate at Indicated Time-points
Description: Respiratory rate of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Breaths per minute
  Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1; Day 1, 1.5 Hours Pre-dose;n=13,13 | 17.2 (2.35) | 16.6 (1.85)
  Period 1;Day 1, 2 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 2 Hours Post-dose;n=13,13 | 15.1 (2.53) | 15.2 (2.09)
  Period 1;Day 1, 4 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 4 Hours Post-dose;n=13,13 | 17.4 (1.89) | 16.5 (2.18)
  Period 1;Day 1, 6 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 6 Hours Post-dose;n=13,13 | 16.6 (1.26) | 16.2 (2.08)
  Period 1;Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 2, 24 Hours Post-dose;n=13,13 | 16.3 (3.15) | 16.6 (2.63)
  Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2; Day 1, 1.5 Hours Pre-dose;n=13,12 | 17.0 (2.16) | 16.7 (1.92)
  Period 2;Day 1, 2 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 2 Hours Post-dose;n=13,12 | 15.0 (2.45) | 16.3 (3.25)
  Period 2;Day 1, 4 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 4 Hours Post-dose;n=13,12 | 15.7 (2.69) | 16.8 (1.59)
  Period 2;Day 1, 6 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 6 Hours Post-dose;n=13,12 | 15.8 (2.51) | 16.2 (2.48)
  Period 2;Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 2, 24 Hours Post-dose;n=13,12 | 16.8 (1.92) | 17.2 (2.48)

24. Secondary Outcome: Pulse Rate at Indicated Time-points
Description: Pulse rate of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Beats per minute
  Period 1;Day 1, 1.5 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 1.5 Hours Pre-dose;n=13,13 | 63.2 (11.29) | 69.4 (12.99)
  Period 1;Day 1, 2 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 2 Hours Post-dose;n=13,13 | 64.2 (9.41) | 67.0 (12.17)
  Period 1;Day 1, 4 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 4 Hours Post-dose;n=13,13 | 65.5 (11.30) | 68.2 (12.75)
  Period 1;Day 1, 6 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 6 Hours Post-dose;n=13,13 | 72.5 (11.83) | 76.6 (13.30)
  Period 1;Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 2, 24 Hours Post-dose;n=13,13 | 63.5 (9.63) | 63.9 (10.67)
  Period 2;Day 1, 1.5 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 1.5 Hours Pre-dose;n=13,12 | 67.4 (13.00) | 66.0 (10.26)
  Period 2;Day 1, 2 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 2 Hours Post-dose;n=13,12 | 67.0 (9.51) | 66.3 (11.36)
  Period 2;Day 1, 4 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 4 Hours Post-dose;n=13,12 | 67.8 (11.26) | 68.8 (10.28)
  Period 2;Day 1, 6 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 6 Hours Post-dose;n=13,12 | 76.8 (11.06) | 78.0 (12.17)
  Period 2;Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 2, 24 Hours Post-dose;n=13,12 | 67.2 (9.07) | 66.3 (10.01)

25. Secondary Outcome: Body Temperature at Indicated Time-points
Description: Body temperature of participants was measured on Day 1 and Day 2 of each treatment period 1 and 2 in a supine position after 5 minutes rest. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 2 of each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
Number analyzed (Participants) | 26 | 25
Degree Celsius
  Period 1;Day 1, 1.5 Hours Pre-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 1.5 Hours Pre-dose;n=13,13 | 36.43 (0.455) | 36.47 (0.440)
  Period 1;Day 1, 2 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 2 Hours Post-dose;n=13,13 | 36.68 (0.393) | 36.62 (0.430)
  Period 1;Day 1, 4 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 4 Hours Post-dose;n=13,13 | 36.51 (0.377) | 36.48 (0.443)
  Period 1;Day 1, 6 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 1, 6 Hours Post-dose;n=13,13 | 36.55 (0.433) | 36.81 (0.403)
  Period 1;Day 2, 24 Hours Post-dose;n=13,13: number analyzed (Participants) | 13 | 13
  Period 1;Day 2, 24 Hours Post-dose;n=13,13 | 36.33 (0.312) | 36.38 (0.363)
  Period 2;Day 1, 1.5 Hours Pre-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 1.5 Hours Pre-dose;n=13,12 | 36.28 (0.396) | 36.14 (0.300)
  Period 2;Day 1, 2 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 2 Hours Post-dose;n=13,12 | 36.62 (0.361) | 36.17 (0.334)
  Period 2;Day 1, 4 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 4 Hours Post-dose;n=13,12 | 36.75 (0.454) | 36.63 (0.234)
  Period 2;Day 1, 6 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 1, 6 Hours Post-dose;n=13,12 | 36.62 (0.392) | 36.75 (0.480)
  Period 2;Day 2, 24 Hours Post-dose;n=13,12: number analyzed (Participants) | 13 | 12
  Period 2;Day 2, 24 Hours Post-dose;n=13,12 | 36.38 (0.458) | 36.38 (0.414)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and Non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to 4 weeks in each treatment period.
Description: SAEs and Non-SAEs were reported by treatment for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment.
Arm/Group | GR37547 500 mg | Ciprofloxacin 500 mg Reference
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 6/26 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GR37547 500 mg (N=26) | Ciprofloxacin 500 mg Reference (N=25)
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 2
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03150082/Prot_SAP_001.pdf